CLINICAL TRIAL: NCT07334886
Title: A Study to Investigate the Absorption, Metabolism, and Excretion of [14C]Ulonivirine in Healthy Adults
Brief Title: A Study of [14C]Ulonivirine ([14C]MK-8507) in Healthy Adults (MK-8507-006)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8507-006; MK-8507-006 (Other: MSD)
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]Ulonivirine (Experimental): All participants receive a single oral dose of [14C]ulonivirine on Day 1.
  Interventions: Drug: [14C]Ulonivirine

INTERVENTIONS:
Drug: [14C]Ulonivirine — Oral Solution
  Other Names: [14C]ULO; [14C]MK-8507

SUMMARY:
The goal of this study is to learn how [14C]ulonivirine moves through a healthy person's body over time. Researchers will study how [14C]ulonivirine is absorbed by the body, broken down by the body, and how it leaves the body.

ELIGIBILITY:
Key Inclusion Criteria include but are not limited to:

* Is in good health
* Has a body mass index (BMI) of 18 to 32 kg/m^2

Key Exclusion Criteria include but are not limited to:

* Has a history of cancer
* Has positive tests for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus antibody

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2025-09-17 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Cumulative Percentage of Total Radioactivity Recovered (FE) from Urine and Feces | At designated timepoints (up to approximately 5 weeks postdose)
  Urine and fecal samples will be collected to determine the cumulative percentage of radioactivity recovered from both urine and feces.
FE from Urine | At designated timepoints (up to approximately 5 weeks postdose)
  Urine samples will be collected to determine the percent of total radioactivity recovered from urine.
FE from Feces | At designated timepoints (up to approximately 5 weeks postdose)
  Fecal samples will be collected to determine the percent of total radioactivity recovered from feces.
Cumulative Amount of Radioactivity Recovered from Urine | At designated timepoints (up to approximately 5 weeks postdose)
  Urine samples will be collected to determine the cumulative amount of radioactivity recovered from urine.
Percent of Total Radioactive Dose Recovered from Urine | At designated timepoints (up to approximately 5 weeks postdose)
  Urine samples will be collected to determine the percent of the total radioactive dose recovered from urine.
Cumulative Amount of Radioactivity Recovered from Feces | At designated timepoints (up to approximately 5 weeks postdose)
  Fecal samples will be collected to determine the cumulative amount of radioactivity recovered from feces.
Percent of Total Radioactive Dose Recovered from Feces | At designated timepoints (up to approximately 5 weeks postdose)
  Fecal samples will be collected to determine the percent of the total radioactive dose recovered from feces.
Plasma Ulonivirine: Area Under the Concentration-Time Curve from Time 0 to Time of the Last Concentration (AUC0-last) | At designated timepoints (up to approximately 2 weeks postdose)
  Plasma samples will be collected to determine the AUC0-last of ulonivirine.
Plasma Ulonivirine: Area Under the Concentration-Time Curve from Time 0 Extrapolated to Infinity (AUC0-inf) | At designated timepoints (up to approximately 2 weeks postdose)
  Plasma samples will be collected to determine the AUC0-inf of ulonivirine.
Plasma Ulonivirine: Maximum Observed Concentration (Cmax) | At designated timepoints (up to approximately 2 weeks postdose)
  Plasma samples will be collected to determine the Cmax of ulonivirine.
Plasma Ulonivirine: Concentration at 168 Hours Postdose (C168) | At approximately 1 week postdose
  Plasma samples will be collected to determine the C168 of ulonivirine.
Plasma Ulonivirine: Terminal Half-life (t1/2) | At designated timepoints (up to approximately 2 weeks postdose)
  Plasma samples will be collected to determine the t1/2 of ulonivirine.
Plasma Ulonivirine: Time of Maximum Observed Concentration (Tmax) | At designated timepoints (up to approximately 2 weeks postdose)
  Plasma samples will be collected to determine the Tmax of ulonivirine.
Ratio of Ulonivirine to Total Plasma Radioactivity: AUC0-last (ulonivirine)/ AUC0-last (total radioactivity) | At designated timepoints (up to approximately 5 weeks postdose)
  Plasma samples will be collected to determine the ratio of ulonivirine to total plasma radioactivity: AUC0-last (ulonivirine)/ AUC0-last (total radioactivity)
Plasma Total Radioactivity: AUC0-last | At designated timepoints (up to approximately 5 weeks postdose)
  Plasma samples will be collected to determine the AUC0-last of total radioactivity.
Plasma Total Radioactivity: AUC0-inf | At designated timepoints (up to approximately 5 weeks postdose)
  Plasma samples will be collected to determine the AUC0-inf of total radioactivity.
Plasma Total Radioactivity: Cmax | At designated timepoints (up to approximately 5 weeks postdose)
  Plasma samples will be collected to determine the Cmax of total radioactivity.
Plasma Total Radioactivity: C168 | At approximately 1 week postdose
  Plasma samples will be collected to determine the C168 of total radioactivity.
Plasma Total Radioactivity: t1/2 | At designated timepoints (up to approximately 5 weeks postdose)
  Plasma samples will be collected to determine the t1/2 of total radioactivity.
Plasma Total Radioactivity: Tmax | At designated timepoints (up to approximately 5 weeks postdose)
  Plasma samples will be collected to determine the Tmax of total radioactivity.
Total Number of Metabolites in Plasma that Represent at least 10% of the Dose of Radioactivity | At designated timepoints (up to approximately 5 weeks postdose)
  Plasma samples will be collected at pre-specified timepoints and used to determine the total number of metabolites that represent at least 10% of the dose of radioactivity. Metabolites will be determined using liquid scintillation and high-resolution mass spectrometry.
Total Number of Metabolites in Urine that Represent at least 10% of the Dose of Radioactivity | At designated timepoints (up to approximately 5 weeks postdose)
  Urine samples will be collected at pre-specified timepoints and used to determine the total number of metabolites that represent at least 10% of the dose of radioactivity. Metabolites will be determined using liquid scintillation and high-resolution mass spectrometry.
Total Number of Metabolites in Feces that Represent at least 10% of the Dose of Radioactivity | At designated timepoints (up to approximately 5 weeks postdose)
  Fecal samples will be collected at pre-specified timepoints and used to determine the total number of metabolites that represent at least 10% of the dose of radioactivity. Metabolites will be determined using liquid scintillation and high-resolution mass spectrometry.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 5 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue the Study Due to an AE | Up to approximately 5 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Fortea CRU Madison (Site 002), Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com